CLINICAL TRIAL: NCT00876629
Title: Renal MR Elastography: Normal Findings and Variability of Stiffness Measurements
Brief Title: Renal Magnetic Resonance (MR) Elastography in Healthy Volunteers
Acronym: MRE_Rénale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr Olivier Rouvière, Hôpital E. Herriot
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008.529
Record Dates: First submitted 2009-03-10; First posted 2009-04-07 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2009-08

CONDITIONS: Healthy
Keywords: MR Elastography; kidney; fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pneumatic Driver — Ten healthy volunteers will undergo MR Elastography using a pneumatic driver connected to a commercially available speaker and the stiffness of the left kidney will be measured.
  The examination will be repeated on the same volunteers at least one month later and the same stiffness measurements will be performed.

SUMMARY:
MR Elastography is a new technique aimed at non-invasively measuring the stiffness of tissues. It has recently given interesting results in the assessment of liver fibrosis.

The objectives of the current study are:

1. to develop an imaging protocol for MR Elastography of the kidneys;
2. To calculate the stiffness of normal kidneys;
3. To evaluate the variability of the measurements of kidney stiffness by repeating the procedure twice on the same volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Signed informed consent form
* Insured by the French Social Security

Exclusion Criteria:

* Pregnancy
* Personal or familial history of kidney disease
* Hypertension
* Diabetes
* Contraindication to MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Normal kidney stiffness (measured from MRE data) | 2 months
Variability of stiffness measurement (on repeat examination) | 2 months

SECONDARY OUTCOMES:
Tolerance of the procedure | 2 months
Percentage of partial and total technical failures | 2 months
Quality criteria of stiffness measurements (area of the ROIs used for measurement, mean induced displacement measured in the ROIs) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rouvière, MD, Principal Investigator — Hôpital E. Herriot
Locations (1):
- Department of Urinary an Vascular Radiology, Hôpital E. Herriot, Lyon, France

REFERENCES:
- [Result] Rouviere O, Souchon R, Pagnoux G, Menager JM, Chapelon JY. Magnetic resonance elastography of the kidneys: feasibility and reproducibility in young healthy adults. J Magn Reson Imaging. 2011 Oct;34(4):880-6. doi: 10.1002/jmri.22670. Epub 2011 Jul 18. PMID 21769970